CLINICAL TRIAL: NCT05192382
Title: A Randomized, Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Paltusotine in Subjects With Non-pharmacologically Treated Acromegaly (PATHFNDR-2)
Brief Title: A Study to Evaluate the Safety and Efficacy of Paltusotine for the Treatment of Acromegaly (PATHFNDR-2)
Acronym: PATHFNDR-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRN00808-08; 2021-001703-32 (EudraCT Number); 2024-511924-15-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-05; First posted 2022-01-14 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Acromegaly
Keywords: Acromegaly; PATHFNDR; Paltusotine; CRN00808
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paltusotine (Experimental)
  Interventions: Drug: Paltusotine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paltusotine — Paltusotine, tablets, once daily by mouth
  Other Names: CRN00808
  Arms: Paltusotine
Drug: Placebo — Placebo, tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
A randomized, placebo-controlled study designed to evaluate the safety and efficacy of paltusotine (formerly CRN00808; an oral selective nonpeptide somatostatin receptor type 2 biased agonist) in subjects with non-pharmacologically treated acromegaly.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years of age
2. Confirmed diagnosis of acromegaly and either medically naïve, not currently treated, or willing to washout during the study screening period.
3. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, or using effective method(s) of birth control
4. Willing to provide signed informed consent

Exclusion Criteria:

1. Pituitary radiation therapy within 3 years of Screening
2. Prior treatment with paltusotine
3. History of ineffective or intolerance to octreotide or lanreotide
4. History or presence of malignancy except adequately treated basal cell and squamous cell carcinomas of the skin within the past 5 years
5. Use of any investigational drug within the past 30 days or 5 half-lives, whichever is longer
6. Known history of HIV, hepatitis B, or active hepatitis C
7. History of alcohol or substance abuse in the past 12 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study
9. Cardiovascular conditions or medications associated with prolonged QT or those which predispose subjects to heart rhythm abnormalities
10. Subjects with symptomatic cholelithiasis
11. Subjects with clinically significant abnormal findings during the Screening Period, or any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the subject's safety or ability to complete the study
12. Subjects currently or previously using pegvisomant or cabergoline (within 16 weeks prior to Screening) or pasireotide LAR (within 24 weeks prior to Screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2028-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (6):
  - Crinetics Study Site, Aurora, Colorado
  - Crinetics Study Site, Boston, Massachusetts
  - Crinetics Study Site, Columbus, Ohio
  - Crinetics Study Site, Portland, Oregon
  - Crinetics Study Site, Philadelphia, Pennsylvania
  - Crinetics Study Site, Pittsburgh, Pennsylvania
- Argentina (4):
  - Crinetics Study Site, CABA, Buenos Aires
  - Crinetics Study Site, Buenos Aires
  - Crinetics Study Site, CABA
  - Crinetics Study Site, Córdoba
- Brazil (7):
  - Crinetics Study Site, Fortaleza, Ceará
  - Crinetics Study Site, Belo Horizonte, Minas Gerais
  - Crinetics Study Site, Curitiba, Paraná
  - Crinetics Study Site, Botucatu, São Paulo
  - Crinetics Study Site, Campinas, São Paulo
  - Crinetics Study Site, Rio de Janeiro
  - Crinetics Study Site, São Paulo
- Crinetics Study Site, Sofia, Bulgaria
- China (10):
  - Crinetics Study Site (b), Beijing, Beijing Municipality
  - Crinetics Study Site, Guangzhou, Guangdong
  - Crinetics Study Site, Shijiazhuang, Hebei
  - Crinetics Study Site, Zhengzhou, Henan
  - Crinetics Study Site, Wuhan, Hubei
  - Crinetics Study Site, Changsha, Hunan
  - Crinetics Study Site, Jinan, Shandong
  - Crinetics Study Site, Xi’an, Shanxi
  - Crinetics Study Site, Chengdu, Sichuan
  - Crinetics Study Site, Hangzhou, Zhejiang
- France (3):
  - Crinetics Study Site, Marseille
  - Crinetics Study Site, Pessac
  - Crinetics Study Site, Toulouse
- Germany (4):
  - Crinetics Study Site, Aachen
  - Crinetics Study Site, Berlin
  - Crinetics Study Site, München
  - Crinetics Study Site, Würzburg
- Greece (3):
  - Crinetics Study Site, Athens
  - Crinetics Study Site (b), Athens
  - Crinetics Study Site, Thessaloniki
- Hungary (2):
  - Crinetics Study Site, Budapest
  - Crinetics Study Site, Pécs
- India (6):
  - Crinetics Study Site, Bangalore, Karnataka
  - Crinetics Study Site, Belagavi, Karnataka
  - Crinetics Study Site, Kochi, Kerala
  - Crinetics Study Site, Mumbai, Maharashtra
  - Crinetics Study Site, Chandigarh
  - Crinetics Study Site, Delhi
- Crinetics Study Site, Petah Tikva, Israel
- Crinetics Study Site, Roma, Italy
- Poland (3):
  - Crinetics Study Site, Bydgoszcz
  - Crinetics Study Site, Poznan
  - Crinetics Study Site, Wroclaw
- Crinetics Study Site, Barcelona, Spain
- Crinetics Study Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study where a total of 209 participants were screened, of which 111 participants were randomized (54 participants in the total paltusotine group and 57 participants in the placebo group) to the randomized control (RC) phase.
Pre-assignment Details: Participants were randomized 1:1 to paltusotine or placebo in the RC phase, stratified by prior treatment (medically naive or previously treated versus washout). Those who completed RC or met rescue criteria entered the open-label extension (OLE). The RC phase is complete; the OLE is ongoing.
Groups:
- RC: Paltusotine Then OLE: Participants were randomized in a 1:1 ratio and received a daily dose of paltusotine orally.
- RC: Placebo Then OLE: Participants were randomized to receive matching placebo tablets in a 1:1 ratio.
- Direct to OLE: Paltusotine: At the completion of study enrollment, participants who met eligibility criteria were directly enrolled in the OLE. The OLE is paltusotine only.
Period: RC Phase (Up to Week 24)
Arm/Group | RC: Paltusotine Then OLE | RC: Placebo Then OLE | Direct to OLE: Paltusotine
Started | 54 | 57 | 0
Completed | 52 | 54 | 0
Not Completed | 2 | 3 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Period: OLE Phase (Up to Week 200)
Arm/Group | RC: Paltusotine Then OLE | RC: Placebo Then OLE | Direct to OLE: Paltusotine
Started | 50 | 52 | 11
Ongoing (OLE is ongoing. Final OLE disposition will be reported after study completion.) | 49 | 48 | 10
Completed | 0 | 0 | 0
Not Completed | 50 | 52 | 11
Not completed — Discontinued | 1 | 4 | 1
Not completed — Ongoing | 49 | 48 | 10

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was the full analysis set (FAS), defined from the intention-to-treat principle and included all randomized subjects. The FAS was the primary analysis set used for efficacy analyses.
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio and received a daily dose of paltusotine orally.
- Placebo: Participants were randomized to receive matching placebo tablets in a 1:1 ratio.
- Total: Total of all reporting groups
Arm/Group | Paltusotine | Placebo | Direct to OLE: Paltusotine | Total
Number analyzed (Participants) | 54 | 57 | 11 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (13.59) | 45.9 (12.30) | 58.4 (8.59) | 50.6 (11.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 33 | 4 | 63
  Male | 28 | 24 | 7 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 18 | 6 | 42
  Not Hispanic or Latino | 31 | 36 | 5 | 72
  Unknown or Not Reported | 5 | 3 | 0 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 15 | 19 | 1 | 35
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 4 | 7
  White | 28 | 30 | 4 | 62
  More than one race | 6 | 4 | 2 | 12
  Unknown or Not Reported | 3 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Biochemical Response in Insulin-like Growth Factor-1 (IGF-1) at the End of the Randomized Control Phase (EOR)
Description: A value >1.0 indicates IGF-1 levels above the age- and sex-adjusted ULN. Response is defined as an IGF-1 level ≤1.0×ULN based on the average of last 2 measurements.
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 54 | 57
percentage of participants | 55.6 | 5.3
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Treatment comparison of all participants receiving paltusotine irrespective of dose levels with Placebo has been presented; Test type: Superiority; p < 0.0001, exact logistic regression model; Odds Ratio (OR) = 42.806, 95% CI 2-sided [8.444 to 455.821]

2. Secondary Outcome: Change in IGF-1 From Baseline to EOT
Description: A value >1.0 indicates IGF-1 levels above the age- and sex-adjusted ULN. Baseline was defined as the last non-missing assessment prior to first dose of study drug for all assessments except IGF-1, growth hormone (GH), and acromegaly symptoms diary (ASD). Change from Baseline was determined by calculating (post-Baseline value - Baseline value).
Time Frame: Baseline to 24 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: nanograms per milliliter (ng/ml)
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 54 | 57
nanograms per milliliter (ng/ml) | -0.819 (0.0789) | 0.087 (0.0751)
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; least square mean difference = -0.906, 95% CI 2-sided [-1.106 to -0.706]

3. Secondary Outcome: Percentage of Participants Achieving IGF-1 <1.3×ULN at EOR
Description: A value >1.0 indicates IGF-1 levels above the age- and sex-adjusted ULN. Response is defined as an IGF-1 level <1.3×ULN based on the average of last 2 measurements.
Time Frame: 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 54 | 57
percentage of participants | 66.7 | 14
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, exact logistic regression model; Odds Ratio (OR) = 18.319, 95% CI 2-sided [5.637 to 79.156]

4. Secondary Outcome: Percentage of Participants With Growth Hormone (GH) Concentration <1 ng/mL at Week 22
Description: The average from integrated GH sampling at week 22 was used to determine response.
Time Frame: Week 22
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 54 | 57
percentage of participants | 57.4 | 17.5
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, exact logistic regression model; Odds Ratio (OR) = 7.588, 95% CI 2-sided [2.776 to 23.483]

5. Secondary Outcome: Change From Baseline in Total Acromegaly Symptoms Diary (ASD) Score to EOT
Description: The ASD is a sponsor-developed daily diary to assess important acromegaly symptoms from the patient perspective. The weekly average ASD total score is calculated from 7 items associated with acromegaly (headache pain, joint pain, sweating, fatigue, weakness in legs, swelling, and numbness or tingling). The ASD total score ranges from 0 to 70 with each symptom contributing up to 10 points. A higher score = higher symptom severity. Change from baseline in total ASD was defined as the postbaseline total ASD score (the average of the available scores seven days on or prior to the scheduled visit date) minus the baseline total ASD score.
Time Frame: Baseline to 24 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Paltusotine | Placebo
Number analyzed (Participants) | 54 | 57
units on a scale | -2.669 (1.4221) | 2.754 (1.3641)
Statistical Analysis 1: Comparison: Paltusotine vs Placebo; Test type: Superiority; p = 0.0039, ANCOVA; least square mean difference = -5.423, 95% CI 2-sided [-9.070 to -1.776]

ADVERSE EVENTS:
Time Frame: Up to 24 weeks
Description: Serious TEAEs and TEAEs were collected in a safety analysis set which was comprised of all participants who received study drug with treatment assignment based on the treatment received. The adverse events are presented as of last participant visit in the RC phase only. Final adverse events from the ongoing OLE will be reported after study completion. All participants, irrespective of their dose level in the paltusotine or placebo arms, have been presented.
Groups:
- Paltusotine: Participants were randomized in a 1:1 ratio and received a daily titrated dose of paltusotine orally.
Arm/Group | Paltusotine | Placebo | Direct to OLE: Paltusotine
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/57 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/57 | 0/11
Other Adverse Events (participants affected / at risk) | 49/54 | 49/57 | 6/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paltusotine (N=54) | Placebo (N=57) | Direct to OLE: Paltusotine (N=11)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paltusotine (N=54) | Placebo (N=57) | Direct to OLE: Paltusotine (N=11)
Diarrhoea (Gastrointestinal disorders) | 18 | 10 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 6 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 10 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 0
Sinusitis (Infections and infestations) | 1 | 4 | 0
Headache (Nervous system disorders) | 11 | 19 | 1
Paraesthesia (Nervous system disorders) | 5 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 13 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 0
Fatigue (General disorders) | 3 | 8 | 1
Peripheral swelling (General disorders) | 2 | 6 | 0
Asthenia (General disorders) | 3 | 3 | 0
Hyperhidrosis (General disorders) | 1 | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 5 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 0
Furuncle (Infections and infestations) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Lipase increased (Investigations) | 2 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 4 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1
Helicobacter test positive (Investigations) | 0 | 0 | 1
Night sweats (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT05192382/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT05192382/SAP_002.pdf